CLINICAL TRIAL: NCT02170974
Title: Bioavailability of BIBR 953 ZW After 150 mg of BIBR 1048 (Oral Pro-drug of BIBR 953 ZW) Administered as HPMC Polymorph II Capsule Relative to 150 mg HPMC Polymorph I Capsule in Healthy Subjects. A Two-way Crossover, Randomised, Open Trial
Brief Title: Bioavailability of BIBR 953 ZW After BIBR 1048 (Oral Pro-drug of BIBR 953 ZW) Administered as Hydroxypropyl Methylcellulose (HPMC) Polymorph II Capsule Relative to HPMC Polymorph I Capsule in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.52
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- BIBR 1048 MS polymorph II (Experimental)
  Interventions: Drug: BIBR 1048 MS polymorph II
- BIBR 1048 MS polymorph I (Active Comparator)
  Interventions: Drug: BIBR 1048 MS polymorph I

INTERVENTIONS:
Drug: BIBR 1048 MS polymorph II
  Arms: BIBR 1048 MS polymorph II
Drug: BIBR 1048 MS polymorph I
  Arms: BIBR 1048 MS polymorph I

SUMMARY:
Investigation of the relative bioavailability of BIBR 953 ZW after administration of 150 mg BIBR 1048 polymorph II versus BIBR 953 ZW after administration of 150 mg BIBR 1048 polymorph I in HPMC capsules

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding at the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation of more than 400 ml within 4 weeks prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the reference range of clinical relevance
* History of any familial bleeding disorder
* Platelets < 150000/μl

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-07; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the plasma concentration-time curve of BIBR 953 ZW from 0 to infinity) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
AUC0-tz | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
Cmax (maximum measured plasma concentration of BIBR 953 ZW) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to when the plasma concentration reaches Cmax after extravascular doses ) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
t1/2 (half life) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
MRTpo (mean time of residence of drug molecules in the body) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
CL/F (apparent clearance after oral administration) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
Vz/F (apparent volume of distribution) | 0 h (predose), 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 24 h, 48 h, and 72 h after drug administration
Changes in ECG | up to 31 days
Changes in systolic and diastolic blood pressure | up to 31 days
Occurrence of adverse events | up to 31 days
Assessment of tolerability by investigator on a four-point scale | up to 31 days